CLINICAL TRIAL: NCT02861937
Title: Estimation of Interleukin-21 Levels in Gingival Crevicular Fluid in Patients With Periodontal Health and Disease Following Non-surgical Periodontal Therapy: A Clinico-biochemical Study
Brief Title: Effect of Non-surgical Periodontal Therapy on Gingival Crevicular Fluid Interleukin-21 Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-D012-36773
Record Dates: First submitted 2016-07-08; First posted 2016-08-10 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Chronic Peridontitis Patients; Chronic Gingivitis; Healthy

STUDY DESIGN:
Intervention Model Description: A total of 34 patients with 19 males and 15 females in the age group of 20-60 years were included. Patients were divided into 3 groups to collect Gingival Crevicular Fluid (GCF) samples for the study.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy (No Intervention): Ten patients with clinically healthy gingiva with probing depth less than 3mm and less than or equal to 10% sites with gingival bleeding on probing present.
  As there was no attachment loss, it was not necessary for us to calculate RAL ( Relative Attachment Level)
- chronic gingivitis (Active Comparator): Chronic gingivitis was defined as having probing depth (PD) less than or equal to 4mm and more than to 25% sites with the gingival bleeding present (BOP)
  As there was no attachment loss, it was not necessary for us to calculate RAL ( Relative Attachment Level)
  Non surgical periodontal therapy (SRP) was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy
  Interventions: Procedure: non surgical periodontal therapy
- chronic periodontitis (Active Comparator): Chronic periodontitis was defined as having probing depth more than or equal to 5mm, RAL more than or equal to 8mm, with more than or equal to 10% sites with BOP positive and evidence of bone loss determined radiographically.
  Non surgical periodontal therapy (SRP) was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy
  Interventions: Procedure: non surgical periodontal therapy

INTERVENTIONS:
Procedure: non surgical periodontal therapy — and root planing (SRP) was performed in two to four appointments lasting approximately 60 minutes each under local anaesthesia (2% lignocaine hydrochloride with 1:2,00,000 adrenaline) using area specific Gracey periodontal curettes and an ultrasonic device. The treatment was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy, which included professional plaque control and reinstruction of oral hygiene.
  Arms: chronic gingivitis; chronic periodontitis

SUMMARY:
Human IL-21 is present in gingival crevicular fluid in periodontal health, gingivitis and chronic periodontitis. A significant increase in the concentration of IL-21 in gingival crevicular fluid is observed with an increase in the amount of periodontal destruction. Non- surgical periodontal therapy aided in decrease of GCF IL-21 levels in clinical gingivitis and chronic periodontitis

DETAILED DESCRIPTION:
Introduction

Periodontal disease is a poly-microbial disease that affects tooth-supporting tissues. Integral part of periodontal disease involves destruction of periodontal tissues that results from stimulation of the bacterial challenge to host immune-inflammatory response. Chronic periodontitis is the most common form of periodontal disease in adult population. The bacterial plaque biofilm is the primitive factor for periodontitis, but the majority of destruction of the periodontal tissues would eventually conclude from a sequence of immune-inflammatory reactions. As a result of cellular activation, inflammatory mediators include cytokines, chemokines etc. collectively contribute to tissue destruction and bone resorption. Cytokines can be grouped as Th1, Th2, Th17 and T regulatory (Treg) based on their expression pattern and effects on target cells or tissues.5 Classically, periodontal disease has been explained by Th1/Th2 pathway. Th1 cells are more frequently detected in the early stage of periodontal lesions suggesting that Th1 cells are associated with a protective response against bacterial infection whereas Th2 cells predominate in the later and advanced period of the disease, having a role in the destruction and progression of periodontal lesions. Alternative type of host response to pathogenic bacteria has been described by the IL-23/IL-17 pathway. This alternative pathway occurs when bacteria induce synthesis of IL-23/17 rather than IL-12, which plays a pivotal role in initiation and maintenance of inflammatory response. IL-23/17 pathway as compared to classical Th1/Th2 pathway is a much fine tuned cellular immune response that has a multitude of functions that bridges the innate and adaptive arm of the immune response.9 Th17 cytokines (IL-17, IL-21, IL-22, IL-6, Tumor necrosis factor {TNF}-a, etc.)8 participate in periodontal disease, but whether their dominant role is host-protective or destructive is questionable. These cytokines have not been elucidated at different inflammatory status in periodontitis.

IL-21 is a type-I cytokine, structurally it appears similar to IL-2, IL-4, and IL-15 proteins. IL-21 is principally composed by activated T cells, but it directs a vast spectrum of myeloid and lymphoid cells of the immune system, which facilitate IL-21 to modulate the acquired and innate immunity.10 IL-21 compete in the immunity against tumor cells11 and chronic viral infections,12 however, enormous accomplishment of IL-21 has been correlated with the advancement of immune inflammatory diseases in various organs.13 IL-21 is heighten in dermatological conditions like skin biopsies14 of patients with systemic lupus erythematosus, psoriasis, and atopic dermatitis. In addition, IL-21 interpretation correspond with the presence of Th17 cells in synovial fluid and peripheral blood of rheumatoid arthritis patients.

Role of IL-21 in inflammation has been extensively studied; the treatment aspect on its levels in periodontal diseases needs to be further explored. Therefore, in the light of the above findings, the investigators determine the levels of interleukin-21 (IL-21) in GCF from chronic gingivitis, chronic periodontitis and control patients before and after non-surgical periodontal therapy along with the co-relation of clinical parameters of periodontal tissues destruction.

MATERIAL AND METHODS:

PATIENTS:

Thirty four patients (19 males and 15 females, aged 20-60 years) were consecutively enrolled over a six month period (April 2014 to September 2014) from the outpatient department of periodontology, Krishnadevaraya College of Dental Sciences, Bangalore, and Karnataka. Ethical clearance for the study was obtained from the institutional ethical committee (02-D012-36773). The study was conducted in accordance with the ethical principles described in the Declaration of Helsinki 2008. Procedure of the study was explained and informed written consent was obtained from all the participants before their inclusion in the study. Among them, 24 patients having diseased periodontium were grouped into 12 chronic gingivitis and 12 chronic periodontitis patients whereas 10 healthy individuals were included as control. Inclusion criteria were: patients having more than or equal to 14 functional teeth, systemically healthy patients who had not received any form of surgical and non surgical periodontal therapy or received antibiotics or non-steroidal anti-inflammatory therapy within the past 6 months of the study. Chronic gingivitis was defined as having probing depth (PD) less than or equal to 4mm and more than to 25% sites with gingival bleeding present (BOP).15 Chronic periodontitis was defined as having probing depth more than or equal to 5mm, RAL more than or equal to 8mm, with more than or equal to 10% sites with BOP positive and evidence of bone loss determined radiographically.16 Patients who volunteered with no evidence of periodontal disease determined by the absence of increased PD or AL were considered as healthy control group.

Clinical Measurements:

Clinical parameters were measured and evaluated for all the teeth excluding 3rd molars, at all the six sites for each tooth (mesio-buccal, disto-buccal, disto-lingual, mid-lingual and mesiolingual). These parameters consisted of pocket depth (PD), assessment of gingival bleeding i.e gingival index (GI), dichotomous measurement of supragingival plaque accumulation i.e plaque index (PI), and bleeding on probing (BOP) to the base of the crevice. One calibrated examiner (MN) performed all the patient evaluations and measurements.

GCF samples collection and analysis:

In all three groups, GCF samples were collected at baseline and 6 weeks post treatment. Site selection was based on the highest score recorded for single site in the oral cavity. A single site in each subject that showed worst inflammatory manifestations (chronic gingivitis) and the highest RAL level (chronic periodontitis) was selected for gingival crevicular fluid collection. In our study, we selected a single site in each subject to avoid pooling of samples from multiple sites, as periodontitis is a site specific disease. Prior to the collection of GCF samples supragingival plaque was removed with cotton pellets avoiding contact with marginal gingiva. Standard paperstrips were carefully inserted to a depth of approximately 2mm, into the sulcus/pocket for 30 seconds for collection of GCF. Blood contaminated strips were discarded and alternative site was used to obtain replacement samples. In chronic gingivitis patients, alternative sample wre collected with the next highest GI scores and in chronic periodontitis patients the next deepest Probing pocket depth {PPD} was selected for the alternative sample site. A calibrated appliance was used to quantify the GCF sample volume and reading were converted to actual volume (μL) by reference to a standard curve, prepared using the periotron reading of volume of fluid (μL) distilled water in perio-col strips. A blank gingival fluid collection (perio-col) strip was placed between the periotron fluid meta sensors and the instrument was adjusted to display a reading of zero. A microlitre syringe was used to accurately deliver 0.25-1.25 μL fluid (distilled water) to perio-col strip. The strips were immediately placed between the periotron sensors. The periotron score volume displayed the known volume of fluid recorded. This step was repeated three more time with 0.25 μL of test fluid and the average score recorded. The above step was repeated using volume of 0.5, 0.75, 1.0, 1.25 μL, and in every instance the mean periotron value calculated and recorded. Once all the score were obtained, a standard curve was computed with known fluid volume (X-axis) and periotron score (Y-axis). In a similar way GCF volumes (from health, chronic gingivitis, chronic periodontitis) from study patients were obtained automatically with periotron score. The interpolation from standard calibration graph gave volume of fluid. After measurement of volume, the strips from the selected sites were placed immediately into individual microcentrifuge tubes containing 200 μL of phosphate buffer solution. The samples were stored at -80 °C until further analysis.

ELISA

The levels of IL-21 in the GCF were determined using ELISA according to the manufactures instruction. To elute the proteins, the tube containing the periopaper strips were vortexed and homogenized for 30 seconds and then centrifuged at 12,500 rpm at 4°C for 5 minutes. The kit used monoclonal antibody MT 21.3 biotin and human recombinant IL-21 standard (captured antibody). Samples were run in triplicate to authenticate the sensitivity of ELISA and all the samples were found to be within the detection limit of ELISA. An ELISA reader (spectramax 190 Ab sorbance microplate reader; molecular devices; Sunnyvale, CA, USA) with 450 nm as elementary wavelength was used to measure the absorbance of the substrate. Conversion of the absorbance readings obtained, into definite volume (pg/mL) were performed using standard reference curve. The protein concentration at each site (pg/mL) were determined by dividing the total amount of IL-21 (pg) by gingival crevicular fluid volume (μL) and subsequently the (pg/μL) values were converted into (pg/mL).

Periodontal treatment protocols:

At baseline, clinical parameters and collection of GCF samples for all patients was done. All patients received a thorough oral hygiene instructions, a full mouth supragingival subgingival scaling along with root planing. Non-surgical periodontal therapy for group III was performed in 2-3 appointments. A single calibrated examiner (MN) provided treatment to all study patients.

STATISTICAL ANALYSIS:

The power of study and sample size calculation was determined on the basis of change in GCF IL-21 level. Current estimates as a pilot study which included 12 patients in each test group and 10 in control group with total sample size of 34 patients. Type II error level of β = 0.20 (80% power) and type I error level of α=0.05 (5% probability) was calculated. The distribution of the samples with respective values of PI, GI, BOP, PD, RAL and IL-21 levels of pre-operatively and post-operatively was analyzed statistically. Data was entered in Microsoft excel and analysed using SPSS {statistical package for social science}, ver.10.05) package. Proportions were compared using Chi-square test (χ2) test of significance. Normality of data was tested using Shapiro-Wilk test. A student t-test was performed to determine pre and post treatment difference values. One way analysis of variance (ANOVA) was used to test the difference between the groups. Comparison of the biochemical and clinical parameters were performed using Kruskal-Wallis non-parametric test. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients having more than or equal to 14 functional teeth, systemically healthy patients who had not received any form of surgical and non surgical periodontal therapy or received antibiotics or non-steroidal anti-inflammatory

Exclusion Criteria:

* smokers pregnant females

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudrakshi Chickanna, MDS, Study Director — Krishnadevaraya college of dental sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty four patients (19 males and 15 females, aged 20-60 years) were consecutively enrolled over a six month period (April 2014 to September 2014) from the outpatient department of periodontology, Krishnadevaraya College of Dental Sciences, Bangalore, and Karnataka.
Pre-assignment Details: 12 chronic gingivitis, 12 chronic periodontitis patients and 10 healthy individuals were included as control. Patients systemically healthy having more than or equal to 14 functional teeth, patients had not received any form of surgical/non surgical periodontal therapy or received antibiotics within the past 6 months.
Groups:
- Group I (Control Group): Healthy: Ten patients with clinically healthy gingiva with probing depth less than 3mm and less than or equal to 10% sites with gingival bleeding on probing present.
- Group II (Test Group I): Chronic Gingivitis: Twelve chronic gingivitis patients having probing depth less than or equal to 4mm and Relative Attachment Level (RAL) less than or equal to 3mm, with more than 25% of sites with gingival bleeding present.
- Group III (Test Group II): Chronic Periodontitis: Twelve chronic periodontitis patients having probing depth more than or equal to 5mm and Relative Attachment Level of more than or equal to 8mm with more than 10% of sites with gingival bleeding on probing present with radiographic evidence of bone loss.
Period: Overall Study
Arm/Group | Group I (Control Group): Healthy | Group II (Test Group I): Chronic Gingivitis | Group III (Test Group II): Chronic Periodontitis
Started | 10 | 12 | 12
Completed | 10 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 34 patients with 19 males and 15 females in the age group of 20-60 years were included. Patients were divided into 3 groups to collect Gingival Crevicular Fluid (GCF) samples for the study.
Groups:
- Group II (Test Group I): Chronic Gingivitis: Chronic gingivitis was defined as having probing depth (PD) less than or equal to 4mm, relative attachment loss (RAL) ) less than or equal to 3mm and more than to 25% sites with gingival bleeding present (BOP)
  Non surgical periodontal therapy (SRP) was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy
  non surgical periodontal therapy: and root planing (SRP) was performed in two to four appointments lasting approximately 60 minutes each under local anaesthesia (2% lignocaine hydrochloride with 1:2,00,000 adrenaline) using area specific Gracey periodontal curettes and an ultrasonic device. The treatment was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy, which included professional plaque control and reinstruction of oral hygiene.
- Group III (Test Group II): Chronic Periodontitis: Chronic periodontitis was defined as having probing depth more than or equal to 5mm, RAL more than or equal to 8mm, with more than or equal to 10% sites with BOP positive and evidence of bone loss determined radiographically.
  Non surgical periodontal therapy (SRP) was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy
  non surgical periodontal therapy: and root planing (SRP) was performed in two to four appointments lasting approximately 60 minutes each under local anaesthesia (2% lignocaine hydrochloride with 1:2,00,000 adrenaline) using area specific Gracey periodontal curettes and an ultrasonic device. The treatment was concluded in 3 weeks. Within the duration of the study, all subjects received supportive therapy, which included professional plaque control and reinstruction of oral hygiene.
- Total: Total of all reporting groups
Arm/Group | Group I (Control Group): Healthy | Group II (Test Group I): Chronic Gingivitis | Group III (Test Group II): Chronic Periodontitis | Total
Number analyzed (Participants) | 10 | 12 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (0.465) | 25 (0.359) | 44 (0.981) | 33 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 15
  Male | 5 | 6 | 8 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 10 | 12 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Pocket Depth
Description: Probing pocket depth (PPD) was recorded using University of North Carolina {UNC}-15 Periodontal probe and customized occlusal stent. Pocket depth was recorded from the crest of the gingival margin to the base of the pocket. The deepest probing pocket depth in the patient"s mouth was considered.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: millimetres
Groups:
- Group I (Control Group): Ten patients with clinically healthy gingiva with probing depth less than 3mm and less than or equal to 10% sites with gingival bleeding on probing present.
- Group II (Test Group I): Twelve chronic gingivitis patients having probing depth less than or equal to 4mm and Relative Attachment Level (RAL) less than or equal to 3mm, with more than 25% of sites with gingival bleeding present.
- Group III (Test Group II): Twelve chronic periodontitis patients having probing depth more than or equal to 5mm and Relative Attachment Level of more than or equal to 8mm with more than 10% of sites with gingival bleeding on probing present with radiographic evidence of bone loss.
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
Number analyzed (Participants) | 10 | 12 | 12
millimetres | 1.60 (0.516) | 2.50 (0.522) | 6.75 (1.138)

2. Primary Outcome: Gingival Index
Description: The severity of Gingivitis was scored on the distolabial papillae, facial margins, mesiolabial papillae and entire lingual gingival margin of each tooth. A blunt instrument such as Periodontal probe was used to assess the bleeding.
  0-Absence of inflammation/normal gingival
  1. Mild inflammation, slight change in color, slight edema; no bleeding on probing
  2. Moderate inflammation; moderate glazing, redness, edema and hypertrophy. Bleeding on probing.The higher the score,worst the outcome
  3. Severe inflammation; marked redness, hypertrophy and ulceration. Tendency to spontaneous bleeding.
  Gingival Score Degree of gingivitis 0.1-1.0-Mild gingivitis 1.1-2.0-Moderate gingivitis 2.1-3.0-Severe gingivitis
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
Number analyzed (Participants) | 10 | 12 | 12
units on a scale | 0.30 (0.041) | 1.71 (0.465) | 2.24 (0.359)

3. Primary Outcome: Plaque Index
Description: The surfaces examined are the four gingival areas of the tooth i,e the distolabial, facial, mesiolabial, and lingual surfaces. Mouth mirror, a light source, a dental explorer, and air drying of the teeth and gingiva were used.
  SCORE CRITERIA 0 No plaque in gingival area
  1. No plaque can be observed by naked eye. A film of plaque adhering to the free gingival margin and adjacent area of the tooth recognized only by running a probe across the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pockets or on the tooth and gingival margin, which can be seen with naked eye.
  3. Abundance of soft matter within the gingival pocket and or on the tooth surface and gingival margin. The interdental area is stuffed with soft debris.
  Plaque Score:Oral Hygiene Status 0:Excellent 0.1-0.9:Good 1.0-1.9:Fair 2.0-3.0:Poor. The higher the value,worst is the outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
Number analyzed (Participants) | 10 | 12 | 12
units on a scale | 0.31 (0.068) | 1.18 (0.597) | 2.14 (0.330)

4. Primary Outcome: Relative Attachment Level:
Description: RAL was measured using UNC-15 periodontal probe and customized acrylic stent. This measurement was made from a fixed reference point from the occlusal surface of the acrylic stent to the base of the periodontal pocket.
  No Relative Attachment Level (RAL) :healthy No Relative Attachment Level (RAL) : chronic gingivitis Relative Attachment Level (RAL) more than or equal to 8mm : chronic periodontitis
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: millimetres
Groups:
- Group II (Test Group I): Twelve chronic gingivitis patients having probing depth less than or equal to 4mm, with no Relative Attachment loss (RAL)and with more than 25% of sites with gingival bleeding present.
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
Number analyzed (Participants) | 10 | 12 | 12
millimetres | 0 (0) | 0 (0) | 9.50 (1.243)

5. Primary Outcome: Interleukin-21(IL-21) Cytokine Levels
Description: IL-21 levels in Gingival crevicular fluid {GCF} was determined by using ELISA kit. Quantikine human IL-21 immunoassay was done according to manufacturer"s instructions (MABTECH SWEDEN)®. ELISA reader was used to record the optical density of the tested samples.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: picogram per millilitres
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
Number analyzed (Participants) | 10 | 12 | 12
picogram per millilitres | 2245.900 (771.718) | 7215.341 (1125.553) | 7390.167 (1982.4)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The Total Number of Participants at Risk equals the number of participants Started in the Participant Flow module, but All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were observed in none.
Arm/Group | Group I (Control Group) | Group II (Test Group I) | Group III (Test Group II)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This study needs to be elucidated with larger sample size and for longer duration, on arresting periodontal disease progression/disease activity by assessing the IL-21 levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No